CLINICAL TRIAL: NCT01492569
Title: Acupuncture Point Stimulation for Treatment of Chemotherapy Nausea and Vomiting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PEDSVAR0016; NCI-2011-03653 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Acute Lymphoblastic Leukemia; Childhood Acute Myeloid Leukemia/Other Myeloid Malignancies; Ewing Sarcoma; Vomiting in Infants and/or Children; Osteosarcoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sarcoma, Ewing; Osteosarcoma | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (TAPS at the P6 point) (Experimental): Patients undergo TAPS at the true acupuncture point (P6) 30 minutes prior to first chemotherapy infusion and then four times a day for 20 minutes every 2 hours at 8am, 10am, 12pm, and 2pm. Patients then crossover to Arm II for the second course of chemotherapy.
  Interventions: Other: questionnaire administration; Procedure: electroacupuncture therapy
- Arm II (TAPS at a non-P6 point) (Sham Comparator): Patients undergo TAPS at a sham non-acupuncture point 30 minutes prior to first chemotherapy infusion and then four times a day for 20 minutes every 2 hours at 8am, 10am, 12pm, and 2pm. Patients then crossover to Arm I for the second course of chemotherapy.
  Interventions: Procedure: electroacupuncture therapy; Other: questionnaire administration

INTERVENTIONS:
Procedure: electroacupuncture therapy — Undergo TAPS at sham point
  Other Names: electroacupuncture
  Arms: Arm II (TAPS at a non-P6 point)
Other: questionnaire administration — Ancillary studies
Procedure: electroacupuncture therapy — Undergo TAPS
  Other Names: electroacupuncture
  Arms: Arm I (TAPS at the P6 point)

SUMMARY:
This randomized pilot clinical trial studies giving acupuncture in reducing nausea and vomiting in patients undergoing chemotherapy. Pressing and stimulating nerves at an acupuncture point on the inside of the wrist may help control nausea and vomiting during chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether transcutaneous acupuncture point stimulation (TAPS) at P6 as an adjuvant treatment to standard antiemetic therapy reduces acute chemotherapy induced nausea and vomiting as compared to sham acupuncture point stimulation in children undergoing their first round of highly or moderately emetogenic chemotherapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo TAPS at the true acupuncture point (P6) 30 minutes prior to first chemotherapy infusion and then four times a day for 20 minutes every 2 hours at 8am, 10am, 12pm, and 2pm. Patients then crossover to Arm II for the second course of chemotherapy.

ARM II: Patients undergo TAPS at a sham non-acupuncture point 30 minutes prior to first chemotherapy infusion and then four times a day for 20 minutes every 2 hours at 8am, 10am, 12pm, and 2pm. Patients then crossover to Arm I for the second course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a planned admission for at least 24 hours for highly emetogenic or moderately emetogenic chemotherapy at Lucile Packard Children's Hospital or Packard El Camino.
* Planned to undergo at least 2 more cycles of chemotherapy.
* Can include but not limited to: children with high risk ALL, AML, Ewing's Sarcoma, Osteosarcoma
* History of vomiting with prior cycles of chemotherapy (2 episodes of emesis at minimum) despite use of conventional antiemetic medications.
* Age 8-21.
* Parent must be able to understand and willing to sign written informed consent document.

Exclusion Criteria:

* Prior knowledge of acupuncture or experience with acupuncture or acupressure.
* There will be no restrictions regarding use of other Investigational Agents.
* Comorbid Diseases:

  * Diagnosis of any cardiac condition (cardiomyopathy, arrhythmia, pacemaker placement).
  * Any diagnosis requiring pediatric intensive care unit admission.
  * Patients with brain tumor, brain metastasis (these patients often require radiation and surgery in addition to chemotherapy which may confound the results)
  * Concomitant radiation therapy during current chemotherapy cycle.
  * Developmental delay patients with allergy to tape or leads will be excluded from the study.
* Pregnant patients will be excluded from the study.
* Cancer survivors will not be excluded from the study as long as they are undergoing chemotherapy treatment for their current cancer therapy.
* HIV-positive patients will not be excluded.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of episodes of vomiting | During the first 24 hours of chemotherapy
Severity of nausea as recorded on the visual analogue scale (VAS) | During the first 24 hours of chemotherapy
  Measured as a continuous variable for the mean episodes of emesis. The mean VAS nausea score will also be measured as a continuous variable. Measured using the Multinational Association of Supportive Care in Cancer (MASCC) antiemesis tool.

SECONDARY OUTCOMES:
Number of as needed (PRN) antiemetic medications needed | After the first 24 hours of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Golianu, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States